CLINICAL TRIAL: NCT00269152
Title: A Randomized Phase 2 Study of Pemetrexed in Combination With Cisplatin or Carboplatin as Adjuvant Chemotherapy in Patients With Completely Resected Stage Ib or II Non-Small Cell Lung Cancer
Brief Title: Feasibility Study of Pemetrexed in Combination With Cisplatin or Carboplatin as Adjuvant Treatment of Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10105; H3E-SB-S089 (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Results first posted 2009-06-11 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Pemetrexed + Cisplatin (Experimental)
  Interventions: Drug: pemetrexed; Drug: cisplatin
- B: Pemetrexed + Carboplatin (Experimental)
  Interventions: Drug: pemetrexed; Drug: carboplatin

INTERVENTIONS:
Drug: pemetrexed — 500 milligrams per square meter (mg/m^2), intravenous (IV), every 21 days x 4 cycles
  Other Names: LY231514; Alimta
Drug: cisplatin — 75 mg/m^2, intravenous (IV), every 21 days x 4 cycles
  Arms: A: Pemetrexed + Cisplatin
Drug: carboplatin — area under the curve (AUC) 5 milligrams per milliliter*minute (mg/ml*min), intravenous (IV), every 21 days x 4 cycles
  Arms: B: Pemetrexed + Carboplatin

SUMMARY:
This study is a multicenter, open-label, two-arm, randomized, parallel Phase 2 feasibility study of pemetrexed in combination with either cisplatin (Arm A) or carboplatin (Arm B) as adjuvant combination-chemotherapy in participants with completely resected, stage Ib or IIa/IIb non-small cell lung cancer (NSCLC).

A two-stage design will be employed independently for both treatment arms, with the possibility of stopping each treatment early for lack of feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non-small cell lung cancer stage Ib, IIa or IIb
* Must have complete tumor resection by pneumonectomy or lobectomy
* Must have been surgically proven to be N2 negative

Exclusion Criteria:

* Serious concomitant systemic disorder
* Post-operative complications or other surgery related conditions
* A prior malignancy other than NSCLC unless that malignancy was diagnosed and treated at least 5 years ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2005-12; Primary Completion 2007-11 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (18):
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Priest-en-Jarez
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Germany (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Berka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bielefeld
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Großhansdorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kassel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Löwenstein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santiago de Compostela

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed + Cisplatin: Pemetrexed: 500 milligrams per square meter (mg/m^2), intravenous (IV), every 21 days x 4 cycles Cisplatin: 75 mg/m^2, intravenous (IV), every 21 days x 4 cycles
- Pemetrexed + Carboplatin: Pemetrexed: 500 mg/m^2, intravenous (IV), every 21 days x 4 cycles Carboplatin: area under the curve (AUC) 5 milligrams per milliliter*minute (mg/ml*min), intravenous (IV), every 21 days x 4 cycles
Period: Overall Study
Arm/Group | Pemetrexed + Cisplatin | Pemetrexed + Carboplatin
Started | 63 (One participant in Pemetrexed+Carboplatin actually received Pemetrexed+Cisplatin) | 59 (4 were randomized without receiving any study drug.)
Completed | 45 | 49
Not Completed | 18 | 10
Not completed — Adverse Event | 9 | 3
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Physician Decision | 2 | 3
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pemetrexed + Cisplatin: Pemetrexed: 500 mg/m^2, intravenous (IV), every 21 days x 4 cycles Cisplatin: 75 mg/m^2, intravenous (IV), every 21 days x 4 cycles
- Pemetrexed + Carboplatin: Pemetrexed: 500 mg/m^2, intravenous (IV), every 21 days x 4 cycles Carboplatin: area under the curve (AUC) 5 mg/ml*min, intravenous (IV), every 21 days x 4 cycles
- Total: Total of all reporting groups
Arm/Group | Pemetrexed + Cisplatin | Pemetrexed + Carboplatin | Total
Number analyzed (Participants) | 63 | 59 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (7.7) | 58.9 (7.2) | 59.7 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 49 | 41 | 90
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 62 | 58 | 120
  African | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  France | 12 | 8 | 20
  Spain | 7 | 8 | 15
  Germany | 44 | 43 | 87
Curative Surgery Used [Number; unit: participants]
  Pneumonectomy | 9 | 9 | 18
  Lobectomy | 46 | 46 | 92
  Bi-lobectomy | 8 | 4 | 12
Smoking History [Number; unit: participants]
  Yes | 56 | 56 | 112
  No | 7 | 3 | 10
Stage of Disease Prior to Tumor Resection [Number; unit: participants] — Classification based on the American Joint Committee on Cancer Staging Criteria for Lung Cancer.
  participants
    Stage Ia | 0 | 1 | 1
    Stage Ib | 27 | 26 | 53
    Stage IIa | 6 | 5 | 11
    Stage IIb | 30 | 25 | 55
    Stage IIIa | 0 | 1 | 1
    Unknown: could have been either Stage IIIb or IV | 0 | 1 | 1
Tumor Type at Initial Pathological Diagnosis [Number; unit: participants]
  Adenocarcinoma of the Lung | 27 | 23 | 50
  Squamous Carcinoma of the Lung | 24 | 20 | 44
  Non-Small Cell Lung Cancer | 5 | 4 | 9
  Mixed Cell (Squamous/Adeno) Carcinoma of Lung | 0 | 5 | 5
  Large Cell Carcinoma of Lung | 5 | 7 | 12
  Bronchoalveolar Carcinoma | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Feasibility of Post-Surgery Chemotherapy
Description: Feasibility was measured by completion of 4 treatment cycles without remaining toxicities >=Grade 3 at 30 days after last infusion.
Time Frame: every 21-day cycle for 4 cycles up to 30 days after last infusion
Population: Number of participants in safety population, that is, number of participants enrolled, randomized and treated with at least one dose of study drug (presented by treatment received arm).
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin | Pemetrexed + Carboplatin
Number analyzed (Participants) | 64 | 54
participants
  Participants "feasible" | 38 | 27
  Non-feasible = Early Discontinuation | 18 | 6
  Non-feasible = Lost to Follow-up | 1 | 2
  Non-feasible = Remaining Grade 3/4 Toxicity | 4 | 3
  Non-feasible = Underdosage (<95% intended dose) | 5 | 19
Statistical Analysis 1: Comparison: Pemetrexed + Cisplatin; Test type: Superiority or Other; Feasibility Response Rate (percentage) = 59.4, 95% CI 2-sided [46.4 to 71.5]
Statistical Analysis 2: Comparison: Pemetrexed + Carboplatin; Test type: Superiority or Other; Feasibility Response Rate (percentage) = 50.0, 95% CI [36.1 to 63.9]

2. Secondary Outcome: Grade III/IV Adverse Events
Description: Number of participants experiencing Grade III/IV hematologic and non-hematologic adverse events possibly related to study drug or protocol procedures in this study.
Time Frame: every 21-day cycle for 4 cycles
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin | Pemetrexed + Carboplatin
Number analyzed (Participants) | 64 | 54
participants
  Neutropenia | 9 | 6
  Anaemia | 0 | 3
  Thrombocytopenia | 0 | 3
  Febrile neutropenia | 0 | 2
  Leukopenia | 0 | 1
  Lymphopenia | 1 | 0
  Neutrophil count decreased | 1 | 6
  Haemoglobin count decreased | 0 | 2
  Platelet count decreased | 1 | 1
  White blood cell count decreased | 0 | 2
  Asthenia | 4 | 2
  Nausea | 3 | 0
  Vomiting | 3 | 0
  Fatigue | 0 | 2
  Catheter related infection | 1 | 0
  Gamma-glutamyltransferase increased | 1 | 0
  Anorexia | 1 | 0
  Hyperglycaemia | 1 | 0
  Hyperkalaemia | 1 | 0
  Psychotic disorder | 1 | 0

3. Secondary Outcome: Overall Survival at 3 Years
Description: For each treatment arm, the Kaplan-Meier technique was used to estimate the 3 year survival rate. Results are presented as probability (%) of survival at 3 years. Overall survival is the duration from enrollment to death. For participants not known to have died, overall survival was censored at the last known alive date.
Time Frame: baseline to date of death from any cause, assessed at 3 years
Population: All randomized participants. Intent to treat population.
Measure: Number (95% Confidence Interval); unit: percent probability of survival (%)
Arm/Group | Pemetrexed + Cisplatin | Pemetrexed + Carboplatin
Number analyzed (Participants) | 63 | 59
percent probability of survival (%) | 82.0 [72.4 to 91.6] | 83.2 [73.2 to 93.2]

4. Secondary Outcome: 3 Year Disease-Free Survival: Probability of Disease-Free Survival at 3 Years
Description: For each treatment arm, the Kaplan-Meier technique was used to estimate the 3 year disease-free rate. Disease-free survival is defined as the time from enrollment to the first observation of disease progression, or death due to any cause. For participants not known to have died and to have had recurrent disease, disease-free survival was censored at the date of the last participant contact with No Recurrence status. Results are presented as probability (%) of disease-free survival at 3 years.
Time Frame: length of time disease free, assessed at 3 years
Population: All randomized participants. Intent to Treat population.
Measure: Number (95% Confidence Interval); unit: probability of disease-free survival (%)
Arm/Group | Pemetrexed + Cisplatin | Pemetrexed + Carboplatin
Number analyzed (Participants) | 63 | 59
probability of disease-free survival (%) | 61.2 [48.3 to 74.0] | 67.3 [54.5 to 80.1]

5. Secondary Outcome: Overall Survival at 6 Years
Description: For each treatment arm, the Kaplan-Meier technique was used to estimate the 6 year survival rate. Results are presented as probability (%) of survival at 6 years. Overall survival is the duration from enrollment to death. For participants not known to have died, overall survival was censored at the last known alive date.
Time Frame: Baseline to date of death from any cause assessed at 6 years
Population: All randomized participants. Intent to treat population.
Measure: Number (95% Confidence Interval); unit: percent probability of survival (%)
Arm/Group | Pemetrexed + Cisplatin | Pemetrexed + Carboplatin
Number analyzed (Participants) | 63 | 59
percent probability of survival (%) | 72.6 [59.3 to 85.9] | 83.2 [73.2 to 93.2]

ADVERSE EVENTS:
Time Frame: baseline through four 21-day cycles and up to 30 days of follow-up after last infusion
Arm/Group | Pemetrexed + Cisplatin | Pemetrexed + Carboplatin
Serious Adverse Events (participants affected / at risk) | 18/64 | 5/54
Other Adverse Events (participants affected / at risk) | 61/64 | 52/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin (N=64) | Pemetrexed + Carboplatin (N=54)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Visual disturbance (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Splenic artery aneurysm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin (N=64) | Pemetrexed + Carboplatin (N=54)
Anaemia (Blood and lymphatic system disorders) | 12 (14) | 8 (9)
Leukopenia (Blood and lymphatic system disorders) | 5 (8) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 21 (34) | 15 (36)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 7 (12)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 3 (3)
Conjunctivitis (Eye disorders) | 1 (1) | 6 (7)
Keratoconjunctivitis sicca (Eye disorders) | 1 (3) | 3 (3)
Lacrimation increased (Eye disorders) | 2 (3) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7) | 5 (6)
Constipation (Gastrointestinal disorders) | 17 (30) | 8 (10)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 7 (11)
Dyspepsia (Gastrointestinal disorders) | 4 (5) | 2 (4)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 40 (82) | 30 (60)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 5 (7)
Vomiting (Gastrointestinal disorders) | 21 (31) | 17 (24)
Asthenia (General disorders) | 10 (22) | 13 (15)
Chest pain (General disorders) | 3 (3) | 4 (6)
Fatigue (General disorders) | 23 (40) | 21 (25)
Mucosal inflammation (General disorders) | 6 (7) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 3 (4)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (5)
Alanine aminotransferase increased (Investigations) | 0 (0) | 6 (8)
Haemoglobin decreased (Investigations) | 2 (2) | 6 (11)
Neutrophil count decreased (Investigations) | 4 (11) | 10 (22)
Platelet count decreased (Investigations) | 4 (9) | 10 (16)
Weight decreased (Investigations) | 3 (5) | 3 (3)
White blood cell count decreased (Investigations) | 2 (4) | 9 (17)
Anorexia (Metabolism and nutrition disorders) | 10 (17) | 14 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5) | 3 (3)
Dysgeusia (Nervous system disorders) | 3 (4) | 7 (9)
Headache (Nervous system disorders) | 8 (12) | 6 (8)
Paraesthesia (Nervous system disorders) | 3 (3) | 4 (4)
Sleep disorder (Psychiatric disorders) | 4 (6) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 16 (19)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 9 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (4)

LIMITATIONS AND CAVEATS:
A protocol amendment was approved after the trial original completed to allow for collection of additional overall survival data due to number of participants surviving at 3 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days